CLINICAL TRIAL: NCT05418296
Title: Assessing a Novel Virtual Environment That Primes Individuals Living With AD/ADRD to Accomplish Activities of Daily Living
Brief Title: Assessing a Novel Virtual Environment That Assists With Activities of Daily Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mandy (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, mandy, Chief Scientific Officer, Mentia DTx
Organization: Mentia DTx (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R43AG071102 (NIH); 1R43AG071102-01A1 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-06-14 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Dementia; Alzheimer Disease; Neurodegenerative Diseases
Keywords: technology; dementia; Alzheimer's disease; virtual; behavioral; cognitive; immersive; caregiver; digital health; videogame; memory; non-pharmacological
MeSH Terms: conditions — Dementia; Alzheimer Disease; Neurodegenerative Diseases; Behavior

STUDY DESIGN:
Intervention Model Description: A Virtual Game Environment as a Behavioral Intervention for Alzheimer Disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Persons residing in long-term care homes (Experimental): Subjects' ADLs are studied with intervention compared to baseline (without intervention).
  Interventions: Device: A novel digital health device

INTERVENTIONS:
Device: A novel digital health device — A videogame-generated virtual world designed for the AD/ADRD care dyad.
  Other Names: DevaWorld

SUMMARY:
This Phase 1 study looks at how a new videogame-based program can help residents and care partners prepare for ADLs in a fun way with minimal risk, potentially reducing escalating problems associated with ADL completions.

DETAILED DESCRIPTION:
Central themes in person-centered care are dignity/respect/choice for the care recipient.

This Phase l clinical study is a minimal risk study that focuses on how the new technology can support and amplify these principles, while assisting care staff.

The investigators will use a novel digital health device developed with user-centered design principles, mirroring a range of evidence-based non-pharmacological interventions for people living with Alzheimer's disease and its related dementias (AD/ADRD). This is a purpose-built virtual world depicting activities of daily living (ADLs). It contains interactive engagement stimuli, including customized digital artifacts that hold meaning to the person.

The investigators hypothesize that undertaking ADL-related virtual activities will support completions of actual ADLs, thereby increasing effectiveness and improving care outcomes.

Aim 1: Feasibility Successful outcomes are >55% participation rate and a statistically significant difference between assessments of participation and non-participation, indicating tolerability and acceptability of routine interventions.

Aim 2: Effectiveness

Successful outcomes are:

* a reduction in ADL-related care challenges compared to baseline
* reduced time spent on the evening ADLs compared to baseline
* a reduction in negative response behaviors associated with the ADL
* greater interest in the ADL
* a positive shift in care staff attitudes

ELIGIBILITY:
Inclusion Criteria:

The subject will have a diagnosis of AD/ADRD, or symptoms of an undiagnosed AD/ADRD as observed by professional care staff and confirmed by the head of clinical care. The investigators will neither include nor exclude participation based on cognitive test scores. The subject will have had challenge(s) completing one or more ADLs in the previous month, as discussed at staff meetings, referenced in care plans, or observed/experienced by direct care staff.

Other specifications:

* Understand English or Russian.
* Can sit comfortably for at least 15 minutes in a chair/wheelchair at a table or propped up in bed or princess chair with a tray table
* Are not known to be in pain
* Have good vision, or good corrected vision (i.e., glasses)
* Have good hearing, or good corrected hearing (i.e., aids)
* May sometimes have anxiety or agitation when undertaking ADLs.

Exclusion Criteria:

Ineligible subjects are those with significant non-AD/ADRD neurological, psychiatric, or physical impairment or those who are totally dependent upon others for ADLs.

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Salomon, PhD, Principal Investigator — Mentia DTx
Locations (2):
- United States (2):
  - Bruceville Point Senior Living Community, Elk Grove, California
  - Elder Ashram, Oakland, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quail Z, Bolton L, Massey K. Digital delivery of non-pharmacological intervention programmes for people living with dementia during the COVID-19 pandemic. BMJ Case Rep. 2021 Jun 17;14(6):e242550. doi: 10.1136/bcr-2021-242550. PMID 34140328
- [Background] Kahle-Wrobleski K, Coley N, Lepage B, Cantet C, Vellas B, Andrieu S; Plasa DSA Group. Understanding the complexities of functional ability in Alzheimer's disease: more than just basic and instrumental factors. Curr Alzheimer Res. 2014 May;11(4):357-66. doi: 10.2174/1567205011666140317101419. PMID 24635843
- [Background] Bourgeois J, Laye M, Lemaire J, Leone E, Deudon A, Darmon N, Giaume C, Lafont V, Brinck-Jensen S, Dechamps A, Konig A, Robert P. Relearning of Activities of Daily Living: A Comparison of the Effectiveness of Three Learning Methods in Patients with Dementia of the Alzheimer Type. J Nutr Health Aging. 2016 Jan;20(1):48-55. doi: 10.1007/s12603-016-0675-4. PMID 26728933
- See also: Database of best dementia care resources — https://bpc.caregiver.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Persons Living With Dementia Residing in Memory Care Communities: Subjects' ADLs are studied with intervention compared to baseline (without intervention).
  A novel digital health device: A videogame-generated virtual world designed for the AD/ADRD care dyad.
- Professional Dementia Caregivers in Memory Care Communities: Subjects are caregivers of the primary participants, ie persons living with dementia
Period: Overall Study
Arm/Group | Persons Living With Dementia Residing in Memory Care Communities | Professional Dementia Caregivers in Memory Care Communities
Started | 28 | 10
Completed | 24 | 9
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Persons Living With Dementia Residing in Memory Care Communities: Subjects' ADLs are studied with intervention compared to baseline (ie., without intervention).
  A novel digital health device: A videogame-generated virtual world designed for the AD/ADRD care dyad.
- Professional Dementia Caregivers in Memory Care Communities: Subjects are the allocated caregivers of the primary participants (i.e., persons living with dementia residing in memory care communities)
- Total: Total of all reporting groups
Arm/Group | Persons Living With Dementia Residing in Memory Care Communities | Professional Dementia Caregivers in Memory Care Communities | Total
Number analyzed (Participants) | 24 | 9 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 9 | 9
  >=65 years | 24 | 0 | 24
Age, Continuous [Mean (Standard Deviation); unit: mean/standard deviation] | 81.1 (8.9) | 36.7 (14.3) | 71.6 (22.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 14 | 0 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 24 | 5 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 4 | 5
  White | 21 | 0 | 21
  More than one race | 0 | 4 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 9 | 33
ADCS-ADL [Mean (Standard Deviation); unit: score on a scale] — Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL- Severe) Collected by survey questionnaire.
  The ADCS-ADL assesses the competence of patients with Alzheimer's Disease (AD) in basic and instrumental activities of daily living (ADLs).Completed by a caregiver in questionnaire format and administered by a clinician/researcher as a structured interview with a caregiver.
  There are 19 questions. The minimum and maximum values are 0 - 54. A higher score means a better outcome. Population: Does not apply to this group
  score on a scale
    number analyzed (Participants) | 16 | 0 | 16
    (all) | 18.9 (8.3) |  | 18.9 (8.3)
NPI-NH [Mean (Standard Deviation); unit: score on a scale] — The Neuropsychiatric Inventory - Nursing Home Version The NPI-NH has been used to characterize the psychopathology of patients in nursing homes as well as to measure the impact of anti dementia and psychotropic drugs and behavioral changes in dementia patients dwelling in nursing homes.
  There are questions. The minimum and maximum values are 12 - 120. A lower score means a better outcome. Administered by a clinician/researcher as a structured interview with a caregiver. Population: Does not apply to this group
  score on a scale
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 20.6 (10.28) |  | 20.6 (10.28)
ADQ [Mean (Standard Deviation); unit: score on a scale] — Approaches to Dementia Questionnaire (ADQ) The ADQ is a validated questionnaire that aims to assess participants' attitudes towards dementia, and has been shown to be reliable, easy to administer and to score. The ADQ is a 19-item survey that assesses attitudes towards people living with dementia using a five-point Likert scale ranging from 'strongly agree' to 'strongly disagree'.
  The total ADQ score ranges from 19 to 95, with higher scores reflecting more positive attitudes towards people living with dementia. Questionnaire completed by caregivers. Population: Does not apply to this group
  score on a scale
    number analyzed (Participants) | 0 | 9 | 9
    (all) |  | 60.2 (2.28) | 60.2 (2.28)
SCIDS [Mean (Standard Deviation); unit: score on a scale] — Sense of Competence in Dementia Care Staff The SCIDS scale provides a useful and user-friendly means of measuring sense of competence in care staff.
  There are questions. The minimum and maximum values are 17 - 68 A higher score means a better outcome. Completed by caregivers Population: Does not apply to this group
  score on a scale
    number analyzed (Participants) | 0 | 9 | 9
    (all) |  | 45.75 (4.09) | 45.75 (4.09)
CBI [Mean (Standard Deviation); unit: score on a scale] — Copenhagen Burnout Inventory(CBI) The (CBI) is a 19-item survey that measures burnout in three areas: personal, work-related, and client-related.
  The total scale ranges from 0 to 300, with high scores indicating high levels of burnout. This inventory is self administered by caregivers. Population: Does not apply to this group
  score on a scale
    number analyzed (Participants) | 0 | 9 | 9
    (all) |  | 116.2 (18.8) | 116.2 (18.8)

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL- Severe)
Description: The ADCS-ADL assesses the competence of patients with Alzheimer's Disease (AD) in basic and instrumental activities of daily living (ADLs). It can be completed by a caregiver in questionnaire format, or administered by a clinician/researcher as a structured interview with a caregiver.
  There are 19 questions. The minimum and maximum values are 0 - 54. A higher score means a better outcome.
Time Frame: 6 weeks
Population: From twenty-four resident participant surveys, eight were excluded from analysis because surveys were a) not filled out or b) incomplete.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Persons Residing in Long-term Care Homes: Participants' ADLs were studied with intervention compared to baseline (without intervention) to identify care dyad acceptance and measure its impact on ADL management.
  Primary participants (memory care residents with AD/ADRD or symptoms of undiagnosed AD/ADRD), across two sites, were introduced to a novel digital health device, "DevaWorld", a videogame-generated virtual home that simulates common ADL activities. The program, which is deployed on touchscreen tablets, contains objects and locations commonly found in the home. Two rooms were selected for the study, a bedroom and a bathroom. A male (Robin) or female (Julie), avatar who reside in the virtual home provided a context for activities, such as "Help Julie clean her teeth" or, "What will Robin wear today?". Graphical 3D objects relevant to the activities under study animate responded to screen taps, and the avatar provided verbal prompts to guide and encourage the participant.
  Participants were supported by an allocated staff- participant recruited to the study. These were regular frontline carers known to the participants who had self-selected for the study from a pool nominated by care team managers. They were formally recruited and underwent training to manage the intervention (both the program and the tablet device on which the program was deployed)
  DevaWorld sessions were run at various times of the day to fit in with staff's daily work flow and availability.
Arm/Group | Persons Residing in Long-term Care Homes
Number analyzed (Participants) | 16
score on a scale | 19.1 (9.9)
Statistical Analysis 1: Comparison: Persons Residing in Long-term Care Homes; Test type: Superiority; p < 0.46, t-test, 1 sided

2. Primary Outcome: The Neuropsychiatric Inventory - Nursing Home Version (NPI-NH) The Minimum and Maximum Values Are A Higher Score Means a Better or Worse Outcome.
Description: The NPI-NH The NPI-NH has been used to characterize the psychopathology of patients in nursing homes as well as to measure the impact of anti dementia and psychotropic drugs and behavioral changes in dementia patients dwelling in nursing homes.
  There are questions. The minimum and maximum values are 12 - 120 A lower score means a better outcome.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persons Living With Dementia Residing in Memory Care Communities
Number analyzed (Participants) | 16
score on a scale | 12.2 (7.6)
Statistical Analysis 1: Comparison: Persons Living With Dementia Residing in Memory Care Communities; Test type: Superiority; p < 0.00314, t-test, 1 sided

3. Secondary Outcome: Approaches to Dementia Questionnaire (ADQ)
Description: The ADQ is a validated questionnaire that aims to assess participants' attitudes towards dementia, and has been shown to be reliable, easy to administer and to score. The ADQ is a 19-item survey that assesses attitudes towards people living with dementia using a five-point Likert scale ranging from 'strongly agree' to 'strongly disagree'.
  The total ADQ score ranges from 19 to 95, with higher scores reflecting more positive attitudes towards people living with dementia.
Time Frame: 6 weeks
Population: All data collected were analysed for five staff participants. Surveys of four were excluded from analysis because surveys were a) not filled out or b) incomplete.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Regular Staff Caregivers of the Primary Participants.: Frontline care staff who had self-selected for the study from a pool nominated by care team managers. They were formally recruited and underwent training to manage the intervention (both the program and the tablet device on which the program was deployed)
  DevaWorld sessions were run at various times of the day to fit in with staff's daily work flow and availability.
Arm/Group | Regular Staff Caregivers of the Primary Participants.
Number analyzed (Participants) | 5
score on a scale | 63.3 (3.21)
Statistical Analysis 1: Comparison: Regular Staff Caregivers of the Primary Participants; Test type: Superiority; p < 0.066, t-test, 1 sided

4. Secondary Outcome: Sense of Competence in Dementia Care Staff (SCIDS) Scale
Description: The SCIDS scale provides a useful and user-friendly means of measuring sense of competence in care staff.
  There are questions. The minimum and maximum values are 17 - 68 A higher score means a better outcome.
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Staff Caregivers of the Primary Participants.
Number analyzed (Participants) | 5
score on a scale | 45.75 (4.08)
Statistical Analysis 1: Comparison: Regular Staff Caregivers of the Primary Participants; Test type: Superiority; p < 0.0850, t-test, 1 sided

5. Secondary Outcome: The Copenhagen Burnout Index
Description: The Copenhagen Burnout Inventory (CBI) is a 19-item survey that measures burnout in three areas: personal, work-related, and client-related.
  Scale ranges from 0 to 300, with high scores indicating high levels of burnout. This inventory is self-administered
Time Frame: 6 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Regular Staff Caregivers of the Primary Participants.
Number analyzed (Participants) | 5
score on a scale | 51.5 (9.23)
Statistical Analysis 1: Comparison: Regular Staff Caregivers of the Primary Participants; Test type: Superiority; p < 0.0716, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: One year
Description: No adverse events
Arm/Group | Persons Living With Dementia Residing in Memory Care Communities | Professional Dementia Caregivers in Memory Care Communities
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/10
Other Adverse Events (participants affected / at risk) | 0/28 | 0/10

LIMITATIONS AND CAVEATS:
Length of study reduced from 8 to 6 weeks due to staff participants' lack of adherence. Reasons: roster changes and absenteeism.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT05418296/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT05418296/ICF_001.pdf